CLINICAL TRIAL: NCT06629285
Title: Effectiveness Comparison Between Continuous Cryotherapy and Ice Pack Therapy After Anterior Cruciate Ligament Reconstruction Surgery
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: University Medical Center Ho Chi Minh City (UMC) (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Supportive Care
Other Study IDs: UMCHoChiMinh
Record Dates: First submitted 2024-10-03; First posted 2024-10-08 (Actual); Last update posted 2024-10-08 (Actual); Status verified 2023-06

CONDITIONS: Postoperative Pain, Acute; Anterior Cruciate Ligament Injuries; Cryotherapy Effect
MeSH Terms: conditions — Pain, Postoperative; Anterior Cruciate Ligament Injuries

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Conventional ice treatment (Active Comparator)
  Interventions: Procedure: Conventional ice treatment
- Continuous compression cryotherapy (Experimental)
  Interventions: Procedure: Continuous compression cryotherapy

INTERVENTIONS:
Procedure: Continuous compression cryotherapy — Using continuous compression cryotherapy around knee after anterior cruciate ligament reconstruction for 3 postoperative days
  Arms: Continuous compression cryotherapy
Procedure: Conventional ice treatment — Using icepack around knee after anterior cruciate ligament reconstruction for 3 postoperative days
  Arms: Conventional ice treatment

SUMMARY:
A randomized controlled trial study conducted by comparing the VAS score, swelling condition, knee ROM and patient's satisfactory score between applying ice pack cold therapy and applying continuous compressive cryotherapy in a postoperative three-day period of anterior cruciate ligament reconstruction surgery patients.

ELIGIBILITY:
Inclusion Criteria:

* Having anterior cruciate ligament reconstruction
* Agree to be enrolled in study

Exclusion Criteria:

* Complex knee injury
* Raynard's disease
* Sensitive to low temperature
* Do not want to use cryotherapy
* Have vascular disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2023-06-01 (Actual); Primary Completion 2024-07-01 (Actual); Study Completion 2024-07-01 (Actual)

PRIMARY OUTCOMES:
Visual Analog Scale | 3 days postoperative
  Compare postoperative Pain score
Knee effusion | 3 days postoperative
  Compare knee swelling rate
Knee range of motion | 3 days postoperative
  Range of motion in knee postoperatively

CONTACTS AND LOCATIONS:
Locations (1):
- University Medical Center, Ho Chi Minh city, Ho Chi Minh City, Ho Chi Minh, Vietnam

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Derived] Tran LTK, Nguyen QTK, Hoang HQ, Nguyen B, Pham VQ. Enhancing patient outcomes after anterior cruciate ligament reconstruction with continuous cryotherapy: A Nursing-Focused Randomized Control Trial. Int J Orthop Trauma Nurs. 2025 Aug;58:101206. doi: 10.1016/j.ijotn.2025.101206. Epub 2025 Jun 11. PMID 40540943